CLINICAL TRIAL: NCT05764278
Title: Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan
Brief Title: The Efficacy and Safety of Early Rehabilitation in Large Vessel Occlusion Patients After Intra-arterial Thrombectomy: A Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111-048-F
Record Dates: First submitted 2022-12-21; First posted 2023-03-10 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Intra-arterial Thrombectomy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effectiveness of earlier rehabilitation intervention after IA thrombectomy(experimental) (Experimental): The effectiveness of early rehabilitation interventions within 24 hours compared with the control group
  Interventions: Other: exercise
- effectiveness of earlier rehabilitation intervention after IA thrombectomy(control) (Active Comparator): The effectiveness of early rehabilitation interventions compared with the experimental group
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — exercise group: first bed exercise after 0~24hr onset ; sit at bed after 24~48hr onset control group: first bed exercise after 24~48hr onset ; sit at bed after 48~72hr onset

SUMMARY:
Early rehabilitation is feasible for stroke patients is still under debate. In addition, IA thrombectomy has been a new treatment for the past few years and currently no known research exploring the efficacy of very early rehabilitation after thrombectomy, or any possible rehabilitation-related adverse effects. Therefore, in this study, the investigators will investigate the effectiveness of earlier rehabilitation intervention after IA thrombectomy for cerebral large vessel occlusion based on functional independence.

DETAILED DESCRIPTION:
The study will be the prospective randomized controlled trial, where patients eligible for inclusion will be randomly assigned to earlier rehabilitation group or control group. The investigators will analyze the correlation between frequency/intensity of rehabilitation and primary/secondary outcomes. Dose-response analysis for earlier rehabilitation will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral stroke due to infarction of large vessels in the anterior circulation, including internal carotid artery (, middle cerebral artery (MCA) M1 or M2 segment, anterior cerebral artery (ACA) A1 segment
2. Receive arterial thrombectomy (IA thrombectomy)
3. Stable vital signs include heartbeat less than 130 bpm, systolic blood pressure less than 180mmHg, blood oxygen SpO2 >92%
4. No use of pressors, oxygen masks or respirators after arterial thrombectomy

Exclusion Criteria:

1. Posterior circulation large vessel stroke
2. Functional score (mRS) ≥ 3 points before the stroke
3. Other contraindications for rehabilitation treatment
4. Neurosurgery immediately after this stroke
5. Those who cannot receive rehabilitation within one week of stroke due to serious medical problems
6. After the stroke, two specialists judged the end of life and arranged palliative and palliative treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 3rd months after stroke
  Modified Rankin Scale (mRS) at 3rd months after stroke:6 grades(higher grades means more disability)

SECONDARY OUTCOMES:
Barthel Index | 1st and 3rd months after stroke
  sum score:0~100(higher score means more functional independence )
Modified Rankin Scale (mRS) | 1st months after stroke
  Modified Rankin Scale (mRS) at 3rd months after stroke:6 grades(higher grades means
Fugl-Meyer Assessment | 1st and 3rd month after stroke
  U/E total score:66 L/E total score:34 the higher score means better movement performance

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch Hsinchu, Taiwan, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No